CLINICAL TRIAL: NCT03642548
Title: A Prospective Multicenter Double-blind Randomized Clinical Trial of Probiotics Combined With Chemotherapy in the Treatment of Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Probiotics Combined With Chemotherapy for Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Ming Li, Associate senior doctor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCCAN
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Probiotics Plus Chemotherapy
Keywords: NSCLC; Bifico; gut-lung axis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A placebo-controlled double-blind randomized study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIFICO Group (Experimental): The intervention group patients receive platinum-based doublet chemotherapy plus BIFICO (Dose: 420mg, 3 times a day, p.o)
  Interventions: Drug: bifico
- Control Gruop (Placebo Comparator): The control group patients receive platinum-based doublet chemotherapy plus Placebo (Dose: 420mg, 3 times a day, p.o)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bifico — Patients in BIFICO group receive platinum-based doublet chemotherapy for first-line treatment chemotherapy plus Bifico.
  Arms: BIFICO Group
Drug: placebo — Patients in control group receive platinum-based doublet chemotherapy for first-line treatment chemotherapy plus Placebo.
  Arms: Control Gruop

SUMMARY:
Based on the theory of intestinal lung axis, the effect of new therapy on patients with advanced NSCLC was observed by adjusting the intestinal micro-ecology and combining existing platinum-based doublet chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary outcomes To compare progression free survival (PFS) and objective response rate (ORR) in patients with stage IIIB or IV non-small cell lung cancer receiving Bifico versus placebo plus platinum-based doublet chemotherapy for first-line treatment.

Secondary outcomes To compare overall survival (OS) between the two arms； To evaluate the nature, severity, and frequency of toxicities between arms； To correlate the blood markers and fecal microbiome (at diagnosis) with outcomes and response.

OUTLINE:

This is a randomized, double-blind, placebo-controlled clinical trial. Patients are stratified according to center, performance status (0 or 1), tobacco use (never vs past or present), weight loss (< 5% vs ≥ 5% or unknown). Patients are randomized to 1 of 2 treatment arms.

BIFICO Group: Patients receive Bifico (420mg, 3 times a day, p.o) plus platinum-based doublet chemotherapy. Chemotherapy repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Placebo Group: Patients receive placebo (420mg, 3 times a day, p.o) plus platinum-based doublet chemotherapy. Chemotherapy repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Blood, tissue and fecal samples are collected and examined for biomarkers, gene mutations and fecal microbiome, and may be banked for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have voluntarily to join the study and give written informed consent for the study.
2. Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic stage IIIB or IV Non-Small Cell Lung Cancer (NSCLC).
3. A cytologic diagnosis is acceptable (i.e., FNA or pleural fluid cytology).
4. Received platinum-based doublet chemotherapy for first-line treatment.
5. At least 1 unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
6. Patients did not receive systemic anti-cancer therapy previously, including traditional Chinese medicine.
7. Able to comply with study and follow-up procedures.
8. Aged 18 to 75 years, ECOG PS: 0~1, estimated survival duration more than 3 months.
9. Major organ function (1) For regular test results (no blood transfusion within 14 days): Hemoglobin（HB）≥90g/L; Absolute neutrophils count（ANC）≥1.5×10^9/L; Blood platelets（PLT）≥80×10^9/L; (2) Biochemical tests results defined as follows: Total bilirubin（TBIL）≤1.5 times the upper limit of normal (ULN); Alanine aminotransferase（ALT）and aspartate amniotransferase AST≤2.5ULNliver metastases if anyALT和AST≤5ULN; Creatinine (Cr)≤1.5ULN or Creatinine Clearance rate (CCr)≥60 ml/min; (3) Patients voluntarily joined the study, signed informed consent, and good compliance.

Exclusion Criteria:

1. Small cell lung cancer (including lung cancer mixed with small cell carcinoma and non-small cell carcinoma).
2. Previously received anti-tumor treatment of any other organs, including radiotherapy, chemotherapy, immunotherapy and Chinese medicine treatment (except for previous radical treatment and no recurrence (treatment of malignant tumor with metastasis time ≥ 5 years).
3. having a variety of factors affecting oral medication (such as inability to swallow, postoperative gastrointestinal resection, chronic diarrhea, intestinal obstruction, etc.).
4. Patients with any severe and/or uncontrolled diseases, such as:

   Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within months prior to randomization, severe uncontrolled arrhythmia; active or uncontrolled serious infections; liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; Active tuberculosis, etc.; uncontrolled hypercalcemia (greater than 1.5 mmol/L calcium or calcium greater than 12 mg/dL or corrected serum calcium greater than ULN), or symptomatic hypercalcemia requiring continued bisphosphonate therapy; Long-term unhealed wounds or fractures.
5. Those who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder.
6. Participated in other clinical trials within four weeks.
7. A history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
8. It is known that there are severe allergic reactions (≥3 grade) to the active ingredients and or any excipients of other test drugs such as pemetrexed, gemcitabine, carboplatin, cisplatin.
9. Use of immunosuppressive drugs within 4 weeks prior to enrollment, excluding nasal glucocorticoids or other routes of topical glucocorticoids or physiological doses of systemic glucocorticoids.
10. known or suspected active autoimmune diseases (congenital or acquired), such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituititis, vasculitis, nephritis, thyroiditis, etc. (Vitiligo or Childhood asthma has been completely relieved, and patients who do not need any intervention after adulthood can be enrolled; patients with well-controlled insulin type I can also be enrolled).
11. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation is known.
12. The history of non-infectious pneumonia requiring glucocorticoid therapy or the current presence of interstitial lung disease in the first year prior to enrollment.
13. Accompanied by other malignant tumors (except for radical treatment, such as cervical carcinoma in situ, non-melanoma skin cancer, etc.); According to the investigator's judgment, there are serious concomitant diseases that endanger the safety of the patient or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-02-21 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 14 months
  Response were evaluated in this study using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee. BEST RESPONSE from the start of study treatment until the end of treatment were reported. Objective response rate is the sum of CR + PR divided by the total number of patients in each group.
Progression Free Survival (PFS) | 6 months
  progression were evaluated using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Randomization to Date of Death from Any Cause.
Number of Participants With Toxicity | up to 12 weeks
  Incidence of Toxicities Measured by NCI CTCAE Version 4.0

REFERENCES:
- [Derived] Xia Q, Chen G, Ren Y, Zheng T, Shen C, Li M, Chen X, Zhai H, Li Z, Xu J, Gu A, Jin M, Fan L. Investigating efficacy of "microbiota modulation of the gut-lung Axis" combined with chemotherapy in patients with advanced NSCLC: study protocol for a multicenter, prospective, double blind, placebo controlled, randomized trial. BMC Cancer. 2021 Jun 22;21(1):721. doi: 10.1186/s12885-021-08448-6. PMID 34157996